CLINICAL TRIAL: NCT06024863
Title: Optimising Screening of Intermediate to High-risk Asymptomatic Sportsmen With Exercise Electrocardiogram. The SEEPRED Study.
Brief Title: Optimising Screening of Intermediate to High-risk Asymptomatic Sportsmen With Exercise Electrocardiogram
Acronym: SEEPRED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN372016/CHUSTE
Record Dates: First submitted 2023-07-27; First posted 2023-09-06 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2022-03

CONDITIONS: Electrocardiography
Keywords: prediction; sport

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sportsmen: Sportsmen (at least 1 hour of physical activity per week) over 35 years of age, referred by their doctor for a screening stress test on a bicycle ergometer in the sports medicine unit from September 2011 to August 2014
  Interventions: Diagnostic Test: Screening stress test on a bicycle ergometer (usual practise)

INTERVENTIONS:
Diagnostic Test: Screening stress test on a bicycle ergometer (usual practise)

SUMMARY:
The importance of exercise electrocardiogram (ECG) is still controversial in the prevention of cardiac events among sportsmen. The aim of this study was to assess the relevance of exercise electrocardiogram (ECG) as a significant prognostic marker for cardiovascular events when any cardiovascular disease (CVD) risk factors are present.

DETAILED DESCRIPTION:
The SEEPRED (Sport, Exercise ECG, prediction) prospective cohort study included leisure time sportsmen over 35 years old who performed exercise electrocardiogram (ECG) screening in the Sports Medicine Unit of the University Hospital of Saint-Etienne from September 2011 to April 2016. Personal, familial history and physical examination were systematically performed before maximal exercise electrocardiogram (ECG). Cardiovascular events and changes in physical activity were searched after exercise electrocardiogram (ECG).

ELIGIBILITY:
Inclusion criteria:

* Patients referred as asymptomatic by their general practitioner for an exercise electrocardiogram (ECG) screening test carried out as a standard procedure for resuming physical activity
* Patients referred as a systematic pre-participation screening to be declared an athlete.

Exclusion criteria:

* Patients with coronary artery disease (CAD) and
* Patients with uninterpretable ST segment due to bundle branch block

Min Age: 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Leisure tim sportmen over 35 years.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Silent Myocardial ischemia (SMI) | Day 1
  Determine the frequency of exercise-induced silent myocardial ischemia (SMI).

SECONDARY OUTCOMES:
Gender record | Day 1
  Gender will be recording during medical consultation in order to predict positive exercise ECG
Age record | Day 1
  Age will be recording during medical consultation in order to predict positive exercise ECG
Physical activity levels record | Day 1
  Physical activity levels will be recording during medical consultation in order to predict positive exercise ECG
Treatment record | Day 1
  Treatment will be recording during medical consultation in order to predict positive exercise ECG
Cardiovascular disease (CVD) risk factors record | Day 1
  Cardiovascular disease (CVD) risk factors will be recording during medical consultation in order to predict positive exercise ECG
Body mass index record | Day 1
  Body mass index will be recording during medical consultation in order to predict positive exercise ECG
Score>5% record | Day 1
  SCORE >5% will be recording during medical consultation in order to predict positive exercise ECG
Maximal heart record | Day 1
  Maximal heart rate will be recording during medical consultation in order to predict positive exercise ECG
Maximal aerobic power record | Day 1
  Maximal aerobic power will be recording during medical consultation in order to predict positive exercise ECG
Maximal blood lactate level record | Day 1
  Maximal blood lactate level will be collected in order to predict positive exercise ECG
Suspected SMI | Day 1
  Exercise ECG screening test
Confirmed SMI | Day 1
  Exercise ECG screening test
Cardiovascular events | Day 1
  Exercise ECG screening test

CONTACTS AND LOCATIONS:
Overall Officials: DAVID HUPIN, MD, Principal Investigator — CHU ST ETIENNE
Locations (1):
- Centre Hospitalier de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hupin D, Oriol M, Laukkanen JA, Abraham P, Dulac N, Laugier S, Trauchessec G, Carmaux A, Haber B, Bertoletti L, Costa AD, Roche F. Screening Sportsmen and Sportswomen Over Age 35: The Relevance of an Exercise Electrocardiogram. Data From the SEEPRED Study. Scand J Med Sci Sports. 2024 Jul;34(7):e14686. doi: 10.1111/sms.14686. PMID 38961532